CLINICAL TRIAL: NCT03331926
Title: Collagenase Clostridium Histolytic is a Common Treatment of MCP and PIP Joint Contractures in Dupuytren Disease. A 1 to 4 Year Followup Study of 198 Joints
Brief Title: Collagenase is a Common Treatment of MCP and PIP Joint Contractures in Dupuytrens Disease
Status: Completed | Type: Observational
Sponsor: Jeppe Lange (Other)
Responsible Party: Sponsor-Investigator, Jeppe Lange, Research secretary, Horsens Hospital
Organization: Horsens Hospital (Other)
Other Study IDs: XIAPEX FOLLOWUP
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Dupuytren Contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — xiapex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Xiapex — Follow-up of effect of treatment

SUMMARY:
To evaluate the effect of collagenase clostridium histolyticum treatment at the Department of Orthopaedic surgery at Horsens Regional Hospital after minimum one-year follow-up (FU).

ELIGIBILITY:
Inclusion Criteria:

* dupuytrens disease
* xiapex treatment

Exclusion Criteria:

- demens/other psychiatric diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who received Xiapex treatment in Horsens from 2013 to May 2016 with a least 1 years of followup.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in extension deficit from baseline to FU in MCP and PIP joints after treatment | Minimum one year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Hartig-Andreasen, MD, PhD, Principal Investigator — Regionshospitalet Horsens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hartig-Andreasen C, Schroll L, Lange J. Clostridium histolyticum as first-line treatment of Dupuytren's disease. Dan Med J. 2019 Feb;66(2):A5527. PMID 30722822